CLINICAL TRIAL: NCT01914237
Title: A Multi-center Trial of Castor Single-Branched Stent Graft System for Endovascular Repair of Aortic Dissection.
Brief Title: A Multi-center Trial of Single-Branched Stent Graft System to Treat Aortic Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Fudan University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Central South University (Other); Beijing Anzhen Hospital (Other); Peking Union Medical College Hospital (Other); Peking University People's Hospital (Other); Chinese PLA General Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Nanjing PLA General Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Shandong Provincial Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other); Xijing Hospital (Other); China Medical University, China (Other); First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Zaiping JING, Director of Department of Vascular Surgery, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Castor-2012-04
Record Dates: First submitted 2013-07-30; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Distal Aortic Dissection
Keywords: Single-Branched Stent Graft System; Aortic Dissection; Endovascular Repair
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Castor Stent Graft (Experimental): To study the safety and efficacy of Castor single-branched stent graft system in endovascular repair of aortic dissection.
  Interventions: Device: Castor Stent Graft

INTERVENTIONS:
Device: Castor Stent Graft — Endovascular Repair of Aortic Dissection
  Other Names: Castor Single-Branched Stent Graft System

SUMMARY:
Aim:Castor is a novel single-branched stent graft system for endovascular repair of aortic arch dissection. This is a prospective, one-arm, open, multi-center, pre-market study of Castor stent to evaluate its efficacy and safety in treatment of aortic dissection.

Number of patients: 70 patients will be included and undertaken endovascular repair with Castor stent.

Follow-up: 1.aortic computed tomographic angiography (CTA) examination 6 and 12 months after the surgery 2.telephone or clinical follow-up 30 days and 2-5 years after the surgery

Primary Outcome Measure: success rate of endovascular repair for efficacy measurement.

Secondary Outcome Measure: 1 year stent related adverse event rate for safety measurement.

Other Outcome Measures:

1. efficacy:

   * 1 year success rate of treatment
   * 1 year patency rate of branch stent
2. safety:

   * in-hospital mortality
   * complication rate of neural system
   * 1 year dissection or stent related mortality

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 80, male or unpregnant female
* diagnosed as aortic dissection
* proximal tear of the dissection locates between 15mm to the distal end of left common carotid artery and 20mm to the distal end of left subclavian artery (LSA) or inverse tear to LSA
* good compliance with the instructions and cooperate with follow-up
* voluntarily signed the informed consent form

Exclusion Criteria:

* Pregnant female
* no appropriate vessel approaches
* patients with connective tissue diseases (such as Marfan syndrome)
* allergic to nitinol or contrast medium
* bad compliance with the instructions and follow-up
* estimated remaining life is less than 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
success rate of endovascular repair | during the surgery
  - during the surgery: successful conduction, accurate positioning and release, and no warping, folding, narrowing or blocking of the stent graft system. Immediately after the stent release, angiography shows both main stent and side arm stent patency, successful exclusion of dissection and no arteriorrhexis or dissection rupture.

SECONDARY OUTCOMES:
1 year stent related adverse event rate | 1 year
  * unexpected breakage and shifting of the stent
  * type I or type III endoleak which needs intervention
  * dissection rupture around the stent

OTHER OUTCOMES:
1 year success rate of treatment | 1 year
  * complete exclusion of the dissection
  * no dissection rupture
  * no type I or type III endoleak which needs twice intervention
  * false lumen of aorta around stent graft closed with thrombus
1 year patency rate of branch stent | 1 year
  The incidence of more than 50% branch stent patency
in-hospital mortality | participants will be followed for the duration of hospital stay, an expected average of 1 week
  mortality of patients caused by dissection related postoperative complications before discharge.
complication rate of neural system | 2 years
  complication rate of neural system related to the stent graft
1 year dissection or stent related mortality | 1 year
  1 year dissection or stent related mortality

CONTACTS AND LOCATIONS:
Overall Officials: Zaiping JING, MD, Principal Investigator — Department of Vascular Surgery, Changhai Hospital
Locations (1):
- Department of Vascular Surgery, Changhai Hospital, Shanghai, Shanghai Municipality, China